CLINICAL TRIAL: NCT03891303
Title: Allogenic Blood Transfusion During Elective Open Abdominal Aortic Surgery and Its Predictors: a Retrospective Database Study at a Tertiary Hospital in Croatia
Brief Title: Allogenic Blood Transfusion During Elective Open Abdominal Aortic Surgery
Status: Completed | Type: Observational
Sponsor: Clinic for Cardiovascular Diseases Magdalena (Network)
Responsible Party: Principal Investigator, Katarina Tomulic Brusich, Principal Investigator, Clinic for Cardiovascular Diseases Magdalena
Other Study IDs: ABT2011-2016
Record Dates: First submitted 2019-03-20; First posted 2019-03-27 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Blood Transfusion
Keywords: Aorta, abdominal; Intraoperative blood salvage; Elective surgical procedures; Patient outcomes assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transfused group (TR): Group received allogenic blood transfusion (ABT) alongside with autologous blood from intraoperative cell saver (ICS) during elective open abdominal aortic surgery.
  Interventions: Other: Allogenic blood transfusion (ABT)
- Non-transfused (non-TR): Group received only autologous blood from intraoperative cell saver (ICS) during elective open abdominal aortic surgery.

INTERVENTIONS:
Other: Allogenic blood transfusion (ABT) — During elective open aortic surgery, the autologous blood from ICS was processed and re-transfused in all patients. However, TR group additionally received ABT.
  Groups: Transfused group (TR)

SUMMARY:
Open surgery on the abdominal aorta is a high risk procedure associated with an intravascular volume blood loss and thereby, with high requirement for blood and blood product transfusion.

The aim of this study was to establish the rate for allogenic blood transfusion (ABT) during elective open abdominal aortic surgery and find parameters associated with ABT requirements.

DETAILED DESCRIPTION:
Two distinct clinical entities affect the abdominal aorta: abdominal aortic aneurysm (AAA) and aortoiliac occlusive disease (AIOD). These are multifactorial vascular disorders caused by complex genetic and environmental factors. Older patients with more comorbidity are often affected. Open abdominal aortic surgery is associated with high mortality rate. Even in specialised institutions it varies from 2 to 5%. Similar results can be compared to mortality for coronary artery bypass grafting. This reflects the complexity of the surgery and the general health of those patients. It is associated with intravascular volume blood loss and, thereby, with a high requirement for blood and blood products transfusion. Allogenic blood transfusion (ABT) has been associated with an increased risk of tumour recurrence, postoperative infection, acute lung injury, perioperative myocardial infarction, postoperative low-output cardiac failure, and increased mortality.

In the last decades, multiple strategies have been undertaken to prevent massive intraoperative blood loss during elective surgery and allogenic blood transfusion requirement. One of the method advocates a preoperative increase in red blood cells level using B12, folic acid and iron supplements or with erythropoietin usage. Other methods involve the optimisation of surgical technique and the use of a machine for intraoperative blood salvage, known as "cell saver".

The aim of this study was to establish the rate for ABT during elective open abdominal aortic surgery, find parameters associated with ABT requirements, and optimise the investigators hospital's maximum surgical blood ordering schedule (MSBOS).

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Elective open abdominal aortic surgery
* Abdominal aortic aneurysm repair
* Abdominal aortic bypass grafting for occlusive aortoiliac disease

Exclusion Criteria:

* Patients younger than 18 years
* Patients undergoing cardiac surgery
* Patients with ruptured abdominal aneurysms
* Patients undergoing endovascular aortic repair
* Patients submitted to other types of vascular surgery (i.e., carotid endarterectomy or peripheral bypass surgery)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A retrospective cross-sectional study was conducted using an existing computerised medical records database at the Department of Anaesthesiology and Intensive Care at the Clinic for Cardiovascular Diseases Magdalena. This Clinic is a tertiary hospital in Croatia specialised in cardiac and vascular surgery. This study is a retrospective analysis of consecutive patients undergoing elective major vascular surgery who had been prospectively risk-stratified.
Sampling Method: Probability Sample
Enrollment: 426 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Overall ABT requirement | Retrospective analysis, 6-year period
  Overall ABT requirement (in %) during elective abdominal aortic surgery with the use of ICS for intraoperative blood salvage and autologous transfusion.

SECONDARY OUTCOMES:
Age as the predictor of higher ABT requirement | Retrospective analysis, 6-year period
  (years)
Gender as the predictors of higher ABT requirement | Retrospective analysis, 6-year period
  male/female
Body mass index (BMI) as the predictors of higher ABT requirement | Retrospective analysis, 6-year period
  BMI (kg/m2)
Body surface area (BSA) as the predictors of higher ABT requirement | Retrospective analysis, 6-year period
  BSA (m²)
Total blood volume as the possible predictors of higher ABT requirement | Retrospective analysis, 6-year period
  TBV (in liters) calculated trough Nadler's formula
Hemoglobin (Hb) and hematocrit (Htc) as the predictors of higher ABT requirement | Retrospective analysis, 6-year period
  Hb (g/L) and Htc (%)
Type of illness as the predictor of higher ABT requirement | Retrospective analysis, 6-year period
  abdominal aortic aneurysm or aortoiliac occlusive disease
Patient's comorbidities as the predictors of higher ABT requirement | Retrospective analysis, 6-year period
  arterial hypertension, coronary artery disease, diabetes, atrial fibrillation, cerebrovascular incidents, chronic obstructive pulmonary disease, chronic renal insufficiency, malignancy
Medications that impair coagulation and homeostasis as the predictor of higher ABT requirement | Retrospective analysis, 6-year period
  acetylsalicylic acid, clopidogrel, or warfarin
Postoperative duration of mechanical ventilation | Retrospective analysis, 6-year period
  (hours)
Length of stay (LOS) | Retrospective analysis, 6-year period
  LOS in ICU (days) and overall hospital LOS (days)
In-hospital mortality rate | Retrospective analysis, 6-year period
  (in %)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kent KC, Zwolak RM, Egorova NN, Riles TS, Manganaro A, Moskowitz AJ, Gelijns AC, Greco G. Analysis of risk factors for abdominal aortic aneurysm in a cohort of more than 3 million individuals. J Vasc Surg. 2010 Sep;52(3):539-48. doi: 10.1016/j.jvs.2010.05.090. Epub 2010 Jul 13. PMID 20630687
- [Background] Ashworth A, Klein AA. Cell salvage as part of a blood conservation strategy in anaesthesia. Br J Anaesth. 2010 Oct;105(4):401-16. doi: 10.1093/bja/aeq244. Epub 2010 Aug 28. PMID 20802228
- [Background] Roubinian NH, Murphy EL, Swain BE, Gardner MN, Liu V, Escobar GJ; NHLBI Recipient Epidemiology and Donor Evaluation Study-III (REDS-III); Northern California Kaiser Permanente DOR Systems Research Initiative. Predicting red blood cell transfusion in hospitalized patients: role of hemoglobin level, comorbidities, and illness severity. BMC Health Serv Res. 2014 May 10;14:213. doi: 10.1186/1472-6963-14-213. PMID 24884605
- [Background] Bursi F, Barbieri A, Politi L, Di Girolamo A, Malagoli A, Grimaldi T, Rumolo A, Busani S, Girardis M, Jaffe AS, Modena MG. Perioperative red blood cell transfusion and outcome in stable patients after elective major vascular surgery. Eur J Vasc Endovasc Surg. 2009 Mar;37(3):311-8. doi: 10.1016/j.ejvs.2008.12.002. Epub 2008 Dec 25. PMID 19111480